## **COVER LETTER**

## Effects of Dry Heat Application on Menstrual Symptoms and Pain:

## **A Randomized Controlled Trial**

Kıvan ÇEVİK KAYA, Dilay AÇIL

Manisa Celal Bayar University, Faculty of Health Sciences, Department of Nursing, Manisa, TURKEY

Mobile: 0(236) 233 09 04

This work was supported by the Manisa Celal Bayar University Scientific Research Projects Coordinator (Project No: 2019-045).

The written informed consents were obtained by participants.

## **Statistical Analysis**

The data of the study were conducted using the Statistical Package for Social Science (SPSS) 23.0 packaged software. In the study, statistical significance difference was calculated on the basis of p<0.05. The students' socio-demographic characteristics and scale-related assessments were performed with the homogeneity test, normality analysis, number and percentage analyses, t-test, variance, and correlation analyses.

Figure-1: CONSORT 2010 Flow Diagram

